CLINICAL TRIAL: NCT00051220
Title: One-Session Treatment for Specific Phobias in Children
Brief Title: Treatment for Specific Phobias in Children
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Virginia Polytechnic Institute and State University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Thomas H. Ollendick, Professor, Virginia Polytechnic Institute and State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R01MH059308 (NIH); R01MH059308 (NIH); DSIR CT-S
Record Dates: First submitted 2003-01-07; First posted 2003-01-08 (Estimated); Last update posted 2013-06-07 (Estimated); Status verified 2013-06

CONDITIONS: Phobic Disorders; Anxiety Disorders
MeSH Terms: conditions — Phobic Disorders; Anxiety Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor

INTERVENTIONS:
Behavioral: One-Session Treatment for Specific Phobias

SUMMARY:
This study will compare the effectiveness of three treatments in reducing symptoms of phobia in children and adolescents.

DETAILED DESCRIPTION:
Children with specific phobias may experience academic, social, and personal distress, as well as interference in day-to-day activities. One-Session Treatment has been found a rapid and effective treatment for adults with phobic disorders. However, its utility in the treatment of childhood phobia has not been examined.

Participants are randomly assigned to 1 of 3 groups: a one-session treatment group, an education/support group, and a waitlist control group. The one-session treatment group is directly exposed to a phobia object or situation during a 3-hour treatment session. In the education/support group, children are given information about fear and phobias and are taught how to deal with them through workbook activities. Children who participate in the one-session treatment group or the education/support group are assessed 1 week post-treatment and again after 6 months. Participants with improved symptoms have a 1-year follow-up. Participants with phobias that persist at 6 months are encouraged to participate in alternative treatment. Waitlist control participants are assessed pre-treatment and 1 month post-treatment. Those who continue to have phobias at the 1-month assessment are randomly assigned to 1 of the 2 active treatments.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of specific phobia disorder

Exclusion Criteria:

* Mental retardation
* Developmental disabilities
* Suicide threat

Ages: 7 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2001-10; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- VA Polytech. Institute and State University, Blacksburg, Virginia, United States
- University of Stockholm, Stockholm, Sweden